CLINICAL TRIAL: NCT07342478
Title: A Phase 3 Open-Label, Randomized, Multicenter Study of Rocbrutinib (LP-168) vs Pirtobrutinib in Covalent BTK Inhibitor (cBTKi) Pretreated Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL) Subjects
Brief Title: ROCKET-CLL Global Phase 3 Study: Rocbrutinib vs Pirtobrutinib in cBTKi-Pretreated R/R CLL/SLL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Newave Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP-168-US-CLL301; ROCKET-CLL (Other: Newave Pharmaceutical Inc.)
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: CLL / SLL; CLL (Chronic Lymphocytic Leukemia); CLL, Refractory; CLL, Relapsed; SLL (Small Lymphocytic Lymphoma); SLL; CLL; CLL Progression
Keywords: Rocbrutinib; LP-168; Pirtobrutinib; Jaypirca; Phase 3; Randomized; Open-label; Relapsed or refractory; CLL; SLL; CLL/SLL; Chronic lymphocytic leukemia; Small lymphocytic lymphoma; Covalent BTK inhibitor pretreated; cBTKi pretreated / cBTKi-exposed; BTK inhibitor; Non-covalent BTK inhibitor; Next-generation BTKi; Dual-binding BTKi; Fourth-generation BTKi; Oral once daily; Progression-free survival; PFS; Independent review committee; IRC-assessed; iwCLL 2018; Lugano 2014; del(17p); TP53 mutation; Prior BCL2 inhibitor exposure; eason for prior BTKi discontinuation (progression vs intolerance); Global
MeSH Terms: conditions — Leukemia, B-Cell; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rocbrutinib (Experimental): 200mg daily
  Interventions: Drug: Rocbrutinib
- Pirtobrutinib (Active Comparator): 200mg daily
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Rocbrutinib — The new generation, highly potent, ultra-selective BTK inhibitor with covalent and non-covalent dual binding mechanism, targeting both WT BTK and mutant BTK
  Arms: Rocbrutinib
Drug: Pirtobrutinib — Pirtobrutinib is a non-covalent BTK inhibitor.
  Arms: Pirtobrutinib

SUMMARY:
This is a Phase 3, randomized, open-label, multicenter study comparing rocbrutinib (LP-168) versus pirtobrutinib in adult participants with relapsed or refractory chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) who have previously received a covalent Bruton's tyrosine kinase inhibitor (cBTKi). Approximately 306 participants will be randomized 1:1 to receive rocbrutinib 200 mg orally once daily or pirtobrutinib 200 mg orally once daily, administered continuously in 28-day cycles until disease progression, unacceptable toxicity, withdrawal of consent, or other discontinuation criteria are met. Randomization will be stratified by presence of del(17p)/TP53 mutation (yes/no), reason for discontinuation of prior cBTKi therapy (toxicity vs disease progression), prior exposure to a BCL2 inhibitor (yes/no), and region (United States/China/rest of world). The primary endpoint is progression-free survival (PFS) assessed by an independent review committee (IRC) using iwCLL 2018 criteria for CLL and Lugano 2014 criteria for SLL. Key secondary objectives include overall survival, overall response rate, time-to-event outcomes, and safety/tolerability; exploratory objectives include health-related quality of life and biomarker assessments.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL) are indolent B-cell malignancies characterized by accumulation of mature but dysfunctional lymphocytes. Covalent Bruton's tyrosine kinase inhibitors (cBTKis) have substantially improved outcomes for patients with CLL/SLL; however, disease progression on cBTKi therapy or intolerance leading to treatment discontinuation remains an important clinical challenge. Patients who discontinue cBTKi therapy due to progression have limited therapeutic options and may experience poor outcomes. Therefore, effective and well-tolerated therapies are needed for participants with relapsed or refractory (R/R) CLL/SLL who have previously received a covalent BTK inhibitor.

Rocbrutinib (LP-168) is a selective next-generation inhibitor of BTK, that can irreversibly inhibit WT BTK, and reversibly inhibit C481 mutated BTK, with activity against known resistance mutations for non-covalent BTKi, under investigation for the treatment of CLL/SLL. Pirtobrutinib is an oral BTK inhibitor with regulatory approval for adults with R/R CLL/SLL who have previously received a covalent BTK inhibitor (cBTKi). This Phase 3 study is designed to compare the efficacy and safety of rocbrutinib versus pirtobrutinib in adult participants with cBTKi-pretreated R/R CLL/SLL.

This is a Phase 3, randomized, open-label, multicenter study conducted at approximately 100 sites globally. Approximately 306 participants will be randomized in a 1:1 ratio to receive rocbrutinib (LP-168) or pirtobrutinib. Eligible participants are adults with confirmed R/R CLL or SLL who require therapy and have received prior treatment with a cBTKi. Participants may have received additional prior systemic therapies, including prior exposure to a BCL2 inhibitor. Key exclusion criteria include central nervous system involvement by CLL/SLL and clinically significant cardiovascular conditions, including uncontrolled arrhythmias and clinically relevant QTc prolongation.

Participants randomized to the investigational arm will receive rocbrutinib 200 mg orally once daily. Participants randomized to the active comparator arm will receive pirtobrutinib 200 mg orally once daily. Study treatments will be administered continuously in 28-day cycles until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-defined discontinuation criteria. Crossover between treatment arms is not permitted.

Randomization will be stratified based on prognostic and treatment-history factors, including: (1) del(17p) and/or TP53 mutation status, (2) reason for discontinuation of prior cBTKi therapy, (3) prior exposure to a BCL2 inhibitor, and (4) geographic region.

The primary endpoint is progression-free survival (PFS). PFS will be assessed by an independent review committee (IRC) to provide objective evaluation of disease status. Response and progression for participants with CLL will be assessed according to iwCLL 2018 criteria, while participants with SLL will be assessed using Lugano 2014 criteria.

Key secondary efficacy endpoints include overall survival (OS), overall response rate (ORR), duration of response (DOR), time to next treatment (TTNT), and event-free survival (EFS). Additional secondary objectives include characterization of the safety and tolerability of rocbrutinib relative to pirtobrutinib. Safety will be assessed through evaluation of adverse events (AEs), serious adverse events (SAEs), adverse events of special interest, deaths, physical examinations, vital signs, electrocardiograms, and clinical laboratory assessments. AEs will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. In addition, population pharmacokinetics will be evaluated to characterize exposure-response relationships.

Exploratory objectives include evaluation of patient-reported outcomes and health-related quality of life, as well as biomarker assessments aimed at characterizing disease biology, mechanisms of response and resistance, and potential predictors of clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Histologically confirmed CLL/SLL iwCLL 2018;
* Relapsed or refractory disease requiring treatment;
* Previously treated with prior lines of therapy including a covalent BTK inhibitor;
* Measurable disease;
* ECOG 0-2;
* Adequate marrow, hepatic, and renal function;
* TP53 mutation status confirmed by NGS;
* 17p deletion status confirmed by FISH;

Exclusion Criteria:

* Prior ncBTKi or BTK degraders;
* Richter's transformation;
* Confirmed prolymphocytic leukemia;
* Uncontrolled comorbidities or infections;
* Known CNS involvement by CLL/SLL;
* Prior malignancy requiring active treatment (except certain adequately treated cancers) per protocol;
* Pregnancy or breastfeeding;
* Concomitant medications or conditions prohibited by protocol (e.g., strong drug-drug interaction risk);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-10-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by IRC | From randomization until disease progression or death from any cause, assessed up to approximately 4 years.
  Progression-Free Survival assessed by independent review committee. PFS is defined as the time from the date of randomization to disease progression or death from any cause, whichever occurs first. Those who do not experience disease progression or death at the time of analysis are censored according to the last evaluation time point.

SECONDARY OUTCOMES:
OS | From randomization until death from any cause, assessed up to approximately 4 years
  Overall survival is defined as the time from the date of randomization to death from any cause. Those who did not die during the analysis were censored according to the last date the subject is known to be alive.
PFS assessed by INV | From randomization until disease progression or death from any cause, assessed up to approximately 4 years.
  Progression free survival assessed by investigator
ORR | From randomization until disease progression, assessed up to approximately 4 years
  Overall response rate
DOR | From first documented response until disease progression or death, assessed up to approximately 4 years
  Duration of response
TTNT | From randomization to start of next anti-CLL/SLL treatment, assessed up to approximately 4 years.
  Time to next treatment
EFS | From randomization until an event occurs, assessed up to approximately 4 years.
  Event free survival
Safety and tolerability | From first dose through 30 days after the last dose of study treatment (up to approximately 4 years)
  Safety and tolerability will be assessed by the incidence, severity, and relationship of adverse events (AEs) and serious adverse events (SAEs), including deaths; adverse events leading to dose modification or discontinuation; and changes in clinical laboratory parameters. Adverse events will be graded per NCI CTCAE v5.0, with specific monitoring for clinically significant cardiac arrhythmias and bleeding events.

OTHER OUTCOMES:
Health related quality of Life | From baseline through end of treatment and follow-up, assessed up to approximately 4 years.
  Health-related quality of life (HRQoL) will be assessed using validated patient-reported outcome (PRO) questionnaires to evaluate participants' functioning and symptoms over time. HRQoL endpoints will include change from baseline in overall health status and selected symptom and function domains. For the Global Health Status/QoL and functional scales, higher scores indicate better quality of life and functioning. For symptom scales/items, higher scores indicate greater symptom burden (worse symptoms).

IPD SHARING:
Plan to Share IPD: Undecided